CLINICAL TRIAL: NCT07214376
Title: A Randomized Placebo-procedure Controlled Trial of the Multi-Pole Pulmonary Artery Radiofrequency Ablation Enhancor System PULmonary Artery Denervation Safety and Efficacy in Patients With Combined Pre- and Post-capillary Pulmonary Hypertension Associated With Left Heart Disease
Brief Title: A Randomized Placebo-procedure Controlled Trial of the Enhancor System (PULmonary Artery Denervation) to Evaluate Safety and Efficacy in Patients With Combined Pre- and Post-capillary Pulmonary Hypertension Associated With Left Heart Disease
Acronym: The PULSE-LHD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pulnovo Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pulnovo-CO-2025-01
Record Dates: First submitted 2025-10-07; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Pulmonary Hypertension; Heart Failure With Reduced Ejection Fraction; Hypertension; Vascular Diseases; Cardiovascular Diseases; Heart Failure; Heart Failure With Preserved Ejection Fraction; Heart Failure With Mid Range Ejection Fraction
Keywords: Pulmonary Artery Denervation; Pulmonary Hypertension Due to Left Heart Disease; Heart Failure; pulmonary hypertension; left heart failure
MeSH Terms: conditions — Hypertension, Pulmonary; Hypertension; Vascular Diseases; Cardiovascular Diseases; Heart Failure

STUDY DESIGN:
Intervention Model Description: At 24 months, control subjects who have experienced a primary efficacy endpoint event and who still meet all eligibility criteria will be offered the opportunity to cross over to the PADN plus GDMT group
Who Masked: Participant, Outcomes Assessor
Masking Description: CEC members
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Pulmonary Artery Denervation (PADN) (Experimental): PADN plus GDMT
  Interventions: Device: Pulmonary Artery Denervation (PADN)
- Control (Active Comparator): Placebo-procedure plus GDMT
  Interventions: Device: Sham procedure control

INTERVENTIONS:
Device: Pulmonary Artery Denervation (PADN) — In patients randomized to Intervention, a Contrast pulmonary artery (PA) angiography will be performed to identify the pulmonary artery bifurcation and measure the PA diameter. Once the anatomy is deemed suitable, a radiofrequency ablation catheter will be introduced into the ostium of the left PA and the distal bifurcation of the main PA. The catheter will be maneuvered within the PA to deliver energy circumferentially, ensuring tight electrode contact with the endovascular surface. Approximately three ablations will be performed at a target temperature of 50 °C (range 45-55 °C) for 120 seconds each at both the left PA ostium and the distal main PA bifurcation.
  All patients enrolled in this clinical study will following the Guideline-Directed Medical Therapy (GDMT)
  Arms: Pulmonary Artery Denervation (PADN)
Device: Sham procedure control — In patients randomized to a placebo-procedure, a script will be followed for approximately 20 minutes to simulate the PADN procedure. All patients enrolled in this clinical study will following the Guideline-Directed Medical Therapy (GDMT)
  Arms: Control

SUMMARY:
The goal of this clinical study is to evaluate the safety and efficacy of percutaneous pulmonary artery denervation with the Multi-Pole Pulmonary Artery Radiofrequency Ablation Enhancor System in patients with combined pre- and post-capillary pulmonary hypertension (CpcPH) associated with left heart disease (LHD). This randomized control trial will compare the investigational device (The Enhancor System) to control (medical therapy.)

Participants who will consist of patients with chronic heart failure (HF) who are receiving maximally tolerated guideline-directed medical therapy (GDMT) for left heart failure, are clinically stable, and who have been diagnosed with CpcPH by right heart catheterization (RHC), will be treated with PADN and followed for 3 years.

DETAILED DESCRIPTION:
Roll-in Subjects:

Prior to enrollment of the first randomized subject at each site, up to two roll-in subjects per operator (maximum 2 operators per site) who meet all eligibility criteria for the randomized trial may be enrolled. Roll-in subjects will receive PADN plus GDMT. Roll-in subjects will undergo all protocol-specified assessments. The sponsor will determine when each operator has achieved acceptable experience with the PADN procedure to advance to the randomized trial, after which no further roll-in patients will be enrolled. Operators who have performed ≥3 prior PADN procedures may not need to enroll a roll-in patient prior to beginning randomization.

Randomized Subjects:

Subjects with CpcPH due to LHD who meet all eligibility criteria will be randomized in a 1:1 ratio (stratified by investigational site and by core laboratory assessed LVEF [≤40% vs >40%]) to one of the two treatment arms:

1. Intervention: PADN plus GDMT
2. Control: Placebo-procedure plus GDMT Subjects will undergo clinical follow-up at 1, 6, 12, 24 and 36 months. At 24 months, control subjects who have experienced a primary efficacy endpoint event and who still meet all eligibility criteria will be offered the opportunity to cross over to the PADN plus GDMT group.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥18 and ≤85 years of age
2. Subject is diagnosed with chronic HF due to left-sided heart disease for at least 6 months prior to screening (regardless of LVEF), and remains symptomatic despite maximally tolerated class I GDMT for left heart failure and CRT as appropriate per US or EU guidelines according to region of enrollment
3. Subject is clinically stable, defined as:

   * No hospitalizations for heart failure for at least 1 month; no major changes in societal guideline-recommended class I oral GDMT for left heart failure for at least 1 month; no CRT or ICD implant in the prior 3 months; and no anticipated major changes in any HF-GDMT (other than possibly diuretic dose) or planned cardiac rhythm management device implantation after the procedure
   * SBP is ≥90 and ≤160 mmHg and resting HR is ≥50 and ≤100 bpm (≤110 bpm for atrial fibrillation)
4. PASP (RVSP) is ≥30 mmHg on the baseline TTE.
5. Subject has New York Heart Association (NYHA) class II, III or IVa symptoms (IVa is defined as symptoms with minimal exertion or at rest, but the patient is able to ambulate and does not require continuous intravenous medications).
6. Subject has 6MWD at baseline ranging from 100 to 450 m limited by dyspnea or fatigue and not orthopedic or other non-HF-related issues
7. Subject has NT-proBNP ≥600 pg/mL for patients with LVEF ≤40% or ≥200 pg/mL for patients with LVEF >40% at the time of screening (a central lab will be made available for sites that cannot measure NT-proBNP)
8. Subject is able and willing to follow all aspects of the research protocol including medication compliance and follow-up visits and testing.
9. Subject or the subject's legally designated representative signs an IRB/EC approved informed consent form prior to study participation.

Exclusion Criteria:

1. Subject has a life expectancy of less than 1 year due to non-cardiovascular causes.
2. Subject has known hypertrophic cardiomyopathy with either left ventricular (LV) outflow tract obstruction or systolic anterior motion (SAM) of the anterior leaflet of the mitral valve; pericardial disease; or infiltrative or active inflammatory myocardial disease, including known amyloidosis
3. Subject has severe stenosis or regurgitation of any heart valve, moderate or severe stenosis of the aortic valve, or any degree of stenosis of the pulmonic valve
4. Subject has symptomatic carotid stenosis, or transient ischemic attack (TIA) or stroke in the prior 30 days or any prior stroke with a permanent residual deficit with modified Rankin Scale (mRS) score ≥4
5. Subject has any prior intracranial hemorrhage with or without a residual deficit, or any known intracranial pathology pre-disposing to bleeding (e.g. mass, AV fistula, aneurysm, etc.)
6. Subjects with a known bleeding diathesis or who will refuse blood transfusions
7. Subjects allergic to heparin (including heparin induced thrombocytopenia), unless bivalirudin or argatroban can be used for procedural anticoagulation
8. Subjects with life threatening allergy to contrast dye that cannot be adequately pre-medicated, or any prior contrast-related anaphylaxis
9. Subject has congenital heart disease other than mitral valve prolapse or a PFO
10. Subject had coronary artery bypass grafting (CABG) or percutaneous coronary intervention (PCI) in the prior 6 months or is anticipated to undergo CABG or PCI within 12 months after randomization.
11. Subject has any pacemaker with an intracardiac sensing or pacing lead or wire implanted in the prior 3 months, or CardioMEMS HF System or other intracardiac pressure monitoring system, or cardiac contractility modulation system or baroreceptor activation therapy implanted within the prior 3 months, or any plans to implant any of these devices within 12 months after the procedure.
12. Subject has undergone atrial fibrillation ablation within the prior 6 months or is anticipated to undergo atrial fibrillation ablation within 12 months after randomization.
13. Subject has undergone heart valve surgery or transcatheter valve intervention within the prior 6 months or is anticipated to undergo heart valve surgery or transcatheter valve intervention (e.g., valve repair or replacement, valvuloplasty) within 12 months after randomization.
14. Subject has any tricuspid or pulmonic valve implants (implanted annuloplasty rings are allowed).
15. Subject has an inferior vena cava (IVC) filter implant.
16. Subject has received a prior heart or heart-lung transplantation or is listed for heart or heart-lung transplantation or is anticipated to receive a ventricular assist device (VAD) implant within 6 months after randomization.
17. Subjects with intracardiac thrombus on TTE.
18. Subjects with pericardial effusion ≥10 mm on TTE
19. Subject's PH is predominantly due to WHO Group 1, 3, 4, or 5. Note: Multifactorial features of PH may be present, but the predominant diagnosis must be WHO Group 2 CpcPH.
20. Subject has been treated with any group 1 PAH-targeted drugs, including sotatercept, within the prior month or is planned to receive such therapy after randomization.
21. Subject is anticipated to undergo any surgery within 6 months after randomization (other than minor surgeries requiring only local anesthesia).
22. Subject has severe renal insufficiency (eGFR <30 mL/min/1.73m2 by the CKD-EPI formula, or on dialysis).
23. Subject has severe liver insufficiency (Child-Pugh classification C).
24. Subject has platelet count <100 × 109/L.
25. Subject has systemic inflammatory or other disease requiring long-term use of oral glucocorticoids or immunosuppressants.
26. Subject has active infection requiring oral or intravenous antibiotics.
27. Subject has a body mass index (BMI) >45 kg/m².
28. Subjects with severe respiratory disease, defined as any disorder of the respiratory system with diffusing capacity of the lungs for carbon monoxide (DLCO) <40% AND total lung capacity (TLC) <60% AND forced expiratory volume in one second (FEV1) <70% by plethysmography; OR who require ambulatory or long-term oxygen therapy
29. Subject has known severe untreated sleep apnea. Note: Subjects with sleep apnea treated with CPAP/BiPAP for at least the prior 3 months are not excluded.
30. Subjects with pulmonary embolism or deep vein thrombosis in the prior 6 months.
31. Subject is a pregnant or breastfeeding woman, or a woman planning to become pregnant within one year. Women of child-bearing potential must have a negative pregnancy test within 1 week of randomization.
32. Subject is participating in another clinical trial of an investigational drug or device that has not reached its primary endpoint.
33. Subject has severe cachexia/frailty, substance abuse, or any other condition that the investigator believes may affect the subject's ability to comply with or complete all the study requirements including follow-up visits.
34. Subject is a member of a vulnerable population who, in the judgment of the investigator, is unable to give Informed Consent for reasons of incapacity, immaturity, adverse personal circumstances or lack of autonomy. This may include individuals with mental disability, children, impoverished persons, persons in prisons, persons in emergency situations, homeless persons, nomads, refugees, and those incapable of giving informed consent. Vulnerable populations may also include members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the Sponsor, members of the armed forces, and persons kept in detention.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint | Immediately after the randomization to last enrolled patient reaches 12-month follow-up
  Composite of Major Heart Failure Events (MHFE). Based on a time-to-first event analysis at 24-month follow-up evaluated when the last enrolled patient reaches 12-month follow-up: 1. Cardiovascular death; 2. Heart transplantation or durable left ventricular assist device (LVAD) implantation; 3.HF hospitalizations; 4. Outpatient worsening HF events
Primary Safety Endpoint | 30-days
  Composite of Device-related or Procedre-related Major Adverse Events (MAEs) in the treatment group compared with a performance goal

SECONDARY OUTCOMES:
Cumulative incidence of Major Heart Failure Events | 30days, 6 months, 12 months, 24 months, and 36 months
  All the following events as following: 1. Cardiovascular death; 2.Heart transplantation or durable left ventricular assist device (LVAD) implantation; 3.HF hospitalizations ; 4.Outpatient worsening HF events
Outpatient worsening HF events | 30days, 6 months, 12 months, 24 months, and 36 months
  Number of outpatients requiring intravenous medication (inotropes, diuretics or vasodilators) due to worsening of heart failure
All cardiovascular hospitalizations | 30days, 6 months, 12 months, 24 months, and 36 months
  Number of patients with cardiovascular hospitalizations
N-terminal pro-B-type natriuretic peptide (NT-proBNP) | 6 months, 12 months, 24 months, and 36 months
  Changes in N-terminal pro-B-type natriuretic peptide (NT-proBNP) from baseline
6 minute walk distance(6MWD) | 6 months, 12 months, 24 months, and 36 months
  6 minute walk distance(6MWD) difference from baseline
Kansas City Cardiomyopathy Questionnaire (KCCQ) | 6 months, 12 months, 24 months, and 36 months
  The KCCQ is a self-administered, questionnaire to provide a better description of quality of life in patients with heart failure. The overall summary score range from 0 to 100, higher score means higher quality of life. Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) overall summary score from baseline to 30 days and 6, 12, 24, and 36 months than baseline
durable left ventricular assist device (LVAD) implantation | 30days, 6 months, 12 months, 24 months, and 36 months
  durable left ventricular assist device (LVAD) implantation (time to first and all events, including recurrent events)
heart transplantation | 30days, 6 months, 12 months, 24 months, and 36 months
  number of heart transplantation (time to first event)
Durable LVAD implantation | 30days, 6 months, 12 months, 24 months, and 36 months
  number of durable LVAD implantation (time to first event)
Cardiovascular death | 30days, 6 months, 12 months, 24 months, and 36 months
  number of cardiovascular death
Atrial septostomy | 30days, 6 months, 12 months, 24 months, and 36 months
  number of atrial septostomy (time to first event)
HF hospitalizations | 30days, 6 months, 12 months, 24 months, and 36 months
  number of HF hospitalizations (time to first and all events, including recurrent events)
Atrial shunt placement | 30days, 6 months, 12 months, 24 months, and 36 months
  Number of atrial shunt placement for all the subjects (time to first event)

OTHER OUTCOMES:
Device-related or Procedure-related Major Adverse Events | 30 days, 6 months, 12 months, 24 months, and 36 months
  Composite of Device-related or Procedure-related Major Adverse Events (MAE) in the treatment group compared with a Performance Goal, defined as the composite of: 1. All-cause mortality; 2.Deep venous thrombosis or pulmonary embolism 3.Perforation or dissection of the pulmonary artery requiring surgical treatment ; 4.Pulmonary artery aneurysm; 5. Pulmonary artery stenosis; 6.Hemoptysis requiring surgical treatment; 7.Left recurrent laryngeal nerve injury; 8. Major vascular complications; 9.BARC type 3 or 5 bleeding; 10.Infection requiring intravenous antibiotics; 11.Endotracheal intubation; 12.Permanent implantation of a pacemaker or defibrillator

CONTACTS AND LOCATIONS:
Overall Officials: Gregg W. Stone, Principal Investigator — Icahn School of Medicine at Mount Sinai

IPD SHARING:
Plan to Share IPD: No